CLINICAL TRIAL: NCT00869713
Title: Long-Term Open-Label Primary Vaccination and Booster Dose Study of the Safety and Immunogenicity of Rift Valley Fever Vaccine, Inactivated, Dried (TSI-GSD 200) in At-Risk Adults
Brief Title: Safety and Immunogenicity Study of Rift Valley Fever Vaccine, Inactivated
Acronym: RVF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: A-15322; FY08-07 (Other: IRB)
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Rift Valley Fever
Keywords: Hemorrhagic Fever; Viral Infections; Neurologic diseases; Arbovirus Infections; RVF
MeSH Terms: conditions — Rift Valley Fever; Hemorrhagic Fevers, Viral; Virus Diseases; Nervous System Diseases; Arbovirus Infections | interventions — Desiccation

STUDY DESIGN:
Intervention Model Description: Open-label, Phase 2, uncontrolled, vaccine study to assess the safety, immunogenicity of RVF (inactivated) vaccine (1.0 mL subcutaneous, SQ).
  Three primary series doses; for responders to the vaccine (PRNT80 ≥ 1:40), 6 month mandatory vaccine booster dose;
  Three primary series doses; for non-responders to the vaccine (PRNT80 < 1:40) may be boosted before 6 months.
Oversight: Data Monitoring Committee: No

ARMS (1):
- primary vaccination with boost (Other): Inactivated, Dried (TSI-GSD 200), RVF Vaccine
  Interventions: Biological: Inactivated, Dried (TSI-GSD 200), RVF Vaccine

INTERVENTIONS:
Biological: Inactivated, Dried (TSI-GSD 200), RVF Vaccine — All subjects: 1.0-mL (SQ)doses on day 0, once between days 7 & 14, & once between days 28-42. Initial responders: A 6-month mandatory vaccine booster dose (1.0 mL, SQ) will be given if the PRNT80 is ≥1:40 after the primary series. Subsequent booster doses will be given for PRNT80 titer <1:40. Initial non-responders: Individual who has a PRNT80 titer <1:40 following the primary series may be administered a booster dose before 6 months. The individual will not receive the mandatory 6-month booster dose. Once an initial non-responder achieves PRNT80 ≥1:40, additional booster doses will be given for subsequent PRNT80 <1:40). All subjects: RVF booster dose will be administered within 90 days after a PRNT80 result of <1:40.

SUMMARY:
This study is designed to determine the safety and immunogenicity of an inactivated Rift Valley Fever (RVF) Vaccine in adults

DETAILED DESCRIPTION:
The primary objectives are to assess safety of Rift Valley Fever (RVF) Vaccine, Inactivated (TSI-GSD 200) and to assess immunogenicity of Rift Valley Fever (RVF) Vaccine, Inactivated (TSI-GSD 200). The secondary objective is to assess incidence of RVF infection in vaccinated personnel

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old.
2. Females of childbearing potential must have a negative serum or urine pregnancy test within 48 hours before each vaccination. Females will be advised not to become pregnant for 3 months after the primary series and each booster dose.
3. Females must not be breast-feeding.
4. Subject must be at risk for exposure to RVF virus.
5. Subject must have an up-to-date (within 1 year) medical history, physical examination, and laboratory tests in their charts and be medically cleared for participation by an investigator. Examinations or tests to qualify for enrollment may be repeated at the discretion of the investigators.
6. Subject must sign and date the approved informed consent document.
7. For initiation of primary series, RVF PRNT80 <1:10.
8. For RE-ENTRY into this protocol or ROLLOVER from an earlier RVF protocol to receive a booster, RVF PRNT80 <1:40 within past 1 year

Exclusion Criteria:

1. Older than 65 years of age for the primary series vaccination (able to receive booster doses if no other contraindications).
2. Clinically significant abnormal lab results, including evidence of Hepatitis C, Hepatitis B carrier state, or elevated (2 times normal) liver function tests.
3. Personal history of immunodeficiency or current treatment with immunosuppressive medication.
4. Confirmed positive human immunodeficiency virus (HIV) titer.
5. Any medical condition that, at the discretion of the physician, may jeopardize the safety of the subject.
6. Any serious or life-threatening allergies to any component of the vaccine: formalin human serum albumin neomycin streptomycin fetal rhesus lung cells RVF virus inactivated
7. Administration of any Investigational New Drug (IND) product or any vaccine within the 28 days before RVF vaccination.
8. Any unresolved adverse event resulting from a previous immunization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
PRNT80 ≥ 1:40 after primary series | Between Days 28-42
  % vaccinated subjects with PRNT80 ≥ 1:40 after primary series (initial responders).
PRNT80 ≥ 1:40 after 6-month mandatory booster dose | 7 months
  % vaccinated subjects with PRNT80 ≥ 1:40 after 6-month mandatory booster dose (initial responders only).
(PRNT80 < 1:40) who responded with a PRNT80 ≥ 1:40 | up to 5 years
  % initial non-responders (PRNT80 < 1:40) who responded with a PRNT80 ≥ 1:40 after 1, 2, 3, or 4 booster doses.
Median duration of PRNT80 ≥ 1:40 in initial responders | up to 5 years
  Median duration of PRNT80 ≥ 1:40 in initial responders after the primary series and 6-month mandatory booster dose.
Median duration of PRNT80 ≥ 1:40 in initial non-responders | up to 5 years
  Median duration of PRNT80 ≥ 1:40 in initial non-responders after the first booster dose that results in PRNT80 ≥ 1:40.
Number of booster doses needed in initial non-responders to achieve PRNT80 ≥ 1:40 | up to 1 year
  Number of booster doses needed in initial non-responders to achieve PRNT80 ≥ 1:40.

SECONDARY OUTCOMES:
Subjects without symptoms | 5 years
  Number of subjects without symptoms
Subjects with any category of local reaction (grade 1-4). | 5 years
  Number of subjects with any local reaction
Subjects with mild, moderate, severe, and potentially life-threatening systemic reactions (grade 1-4). | 5 years
  Number of subjects with systemic reactions
Subjects with generalized allergic reactions | 5 years
  Number of subjects with generalized allergic reactions

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Reisler, MD, Principal Investigator — USAMRIID Medical Division
Locations (1):
- U.S. Army Medical Research Institute of Infectious Diseases, Fort Deterick, Maryland, United States